CLINICAL TRIAL: NCT02613949
Title: A Double-Blinded, Randomized, Sham-Controlled, Study of the Revised NeuroPoint Device for the Treatment of Pain Associated With Fibromyalgia
Brief Title: Prospective Evaluation of RINCE to Reduce Fibromyalgia Effects - 202
Acronym: PERRFECT-202
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cerephex Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NPT-202
Record Dates: First submitted 2015-11-23; First posted 2015-11-25 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; pain; stimulation
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 12-week RINCE mode 1 (Active Comparator): RINCE - active RINCE therapy involving 24 total treatment applications from NeuroPoint device at treatment mode 1
  Interventions: Device: RINCE
- 12-week RINCE mode 2 (Active Comparator): RINCE - active RINCE therapy involving 24 total treatment applications from NeuroPoint device at treatment mode 2
  Interventions: Device: RINCE
- Sham RINCE (Sham Comparator): Sham RINCE - sham RINCE therapy involving 24 total sham applications from NeuroPoint device
  Interventions: Device: RINCE

INTERVENTIONS:
Device: RINCE — The NeuroPoint device is used to deliver repeat applications of RINCE therapy
  Other Names: RINCE therapy; RINCE therapy delivered by the NeuroPoint device

SUMMARY:
The purpose of this study is to test the safety and efficacy of a noninvasive cortical electrostimulation therapy known as "Reduced Impedance Noninvasive Cortical Electrostimulation" (RINCE) in the treatment of pain associated with fibromyalgia. Patients who meet the 2010 American College of Rheumatology criteria for fibromyalgia will receive up to 24 RINCE treatments delivered by a medical device called "NeuroPoint". Approximately 45 fibromyalgia patients will be randomized into one of three study groups. One of these groups will receive sham treatment, meaning they will receive no treatment at all. A second group will receive active RINCE treatment at a nominal signal amplitude level (treatment mode 1). A third group will receive active RINCE treatment at a higher than nominal signal amplitude level (treatment mode 2). The study's primary outcome measure will be the difference between active and sham treatment groups in the mean change from baseline in patients' 24-hour recall average pain scores. The study's hypothesis is that there will be a difference between treatment groups in primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female, 22 to 75 years of age, inclusive.
* Patient has a diagnosis of primary fibromyalgia as defined by the 2010 American College of Rheumatology Preliminary Diagnostic Criteria for fibromyalgia.
* At screening, the patient scores between 40 and 90 on a visual analog scale 24-hour recall pain scale, and between 4 and 9 inclusive on an 11 point numerical rating scale.
* If female, is either not of childbearing potential or is willing to utilize specified practices throughout the study to prevent becoming pregnant.
* Patient is willing and able to refrain or withdraw from the following therapies for the duration of the study: duloxetine, milnacipran, pregabalin, gabapentin, naltrexone, sodium oxybate, and opiates.
* Qualified patients with mild or moderate depression must be clinically stable, without risk of suicidal ideation or behavior, and the dose of allowed anti-depressants should have been stable for at least three months prior to the Baseline clinic visit.
* Patient is willing and able to comply with all protocol-specified requirements.
* Patient is capable of reading and understanding English and has provided written informed consent to participate.

Exclusion Criteria:

* The patient suffers from one or more of clinically significant psychiatric condition that could interfere with the patient's well-being or ability to comply with the protocol.
* Patient has a Beck Depression Inventory-II total score greater than 25 at either the Screening visit or Baseline clinic visit.
* The patient is at increased risk of suicide.
* Patient is unable, unwilling or not advised to refrain from or discontinue prohibited medications or treatments.
* Patient has a diagnosis of, or is being treated for, systemic lupus erythematosus, inflammatory arthritis, or other documented systemic autoimmune disorder, Parkinson's disease, multiple sclerosis, or cancer (other than basal or squamous cell skin cancer).
* Patient has any other chronic pain condition that, in the Investigator's or Sponsor's opinion, could interfere with the patient's assessment of his/her fibromyalgia status.
* Patient has a history of severe, refractory or uncontrolled migraine headaches, seizure disorder or clinically significant cognitive dysfunction.
* Patient is pregnant or planning to become pregnant within the next 6 months.
* Patient has a body mass index greater than 45 at the Screening visit.
* Patient meets any of the study's exclusionary laboratory criteria.
* Patient has any other disease or medical condition that, in the opinion of the Investigator or Sponsor, could endanger the patient, interfere with the evaluation of the study device's efficacy or safety, or compromise the patient's ability to comply with/complete the study.
* Patient has a history of cranial electrical stimulation or transcutaneous magnetic stimulation within 2 years of screening, or electroconvulsive therapy within 5 years of screening; patient was enrolled in the Sponsor's previous NPT-301 study and received greater than 12 stimulation treatments.
* Patient has a metal implant at or above the level of the 7th cervical vertebra, a cardiac pacemaker or defibrillator, or vagus nerve stimulator.
* Any recent surgery or anticipated need for surgery that might confound results or interfere with patient's ability to comply with the protocol.
* Myocardial infarction during the 12 months prior to screening, uncontrolled hypertension, active cardiac disease, clinically significant cardiac rhythm or conduction abnormality, or anticipation of bypass or other cardiac surgery within the next 12 months.
* Current systemic infection (e.g., HIV, hepatitis B or C; Lyme disease).
* Patient is receiving systemic corticosteroids greater than 5 mg prednisone or equivalent per day.
* Patient is using opiates on a regular or frequent basis.
* Pending or current litigation or disability claim (including Workman's Compensation).
* History of significant alcohol and/or drug abuse or dependency within preceding 5 years, or a positive result on the screening (or subsequent) drug screen indicating use of an illicit substance.
* Patient has participated in an investigational study of a therapeutic treatment within 90 days prior to Screening visit or is currently participating in another clinical trial.
* Patient is a staff member or relative of a staff member at either the investigative site or the sponsor.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-11; Primary Completion 2016-07-08 (Actual); Study Completion 2016-07-29 (Actual)

PRIMARY OUTCOMES:
Change from baseline in patients' 24-hour recall average pain intensity | Assessed at 12 weeks
  The primary efficacy endpoint will be the contrast at 12 weeks versus Baseline in the (paired) mean weekly change in patients' self-reported daily (24-hour) recall average pain intensity using an 11-point (0-10) numerical rating scale.

SECONDARY OUTCOMES:
Patient self-reported Global Impression of Change | Assessed at 12 weeks
Change from baseline in Revised Fibromyalgia Impact Questionnaire | Assessed at 12 weeks
Change from baseline in patients' 7 day recall average pain intensity | Assessed at 12 weeks
  Average pain intensity evaluated using an 11-point (0-10) numerical rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: R. Michael Gendreau, MD PhD, Study Director — Cerephex Corporation
Locations (4):
- United States (4):
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Superior Research LLC, Sacramento, California
  - Chicago Research Center, Chicago, Illinois
  - Upstate Clinical Research Associates, Williamsville, New York

REFERENCES:
- [Background] Hargrove JB, Bennett RM, Simons DG, Smith SJ, Nagpal S, Deering DE. A randomized placebo-controlled study of noninvasive cortical electrostimulation in the treatment of fibromyalgia patients. Pain Med. 2012 Jan;13(1):115-24. doi: 10.1111/j.1526-4637.2011.01292.x. PMID 22233397
- [Background] Hargrove JB, Bennett RM, Clauw DJ. Long-term outcomes in fibromyalgia patients treated with noninvasive cortical electrostimulation. Arch Phys Med Rehabil. 2012 Oct;93(10):1868-71. doi: 10.1016/j.apmr.2012.04.006. Epub 2012 Apr 21. PMID 22525670